CLINICAL TRIAL: NCT00861341
Title: Effects of Pioglitazone on Platelet Function
Acronym: UHEM08014
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Charles Francis, Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 24695
Record Dates: First submitted 2009-03-09; First posted 2009-03-13 (Estimated); Results first posted 2016-02-03 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2015-12

CONDITIONS: Diabetes; Platelet Function; Healthy
Keywords: Pioglitazone; Thiazolidinediones; Platelet Function; Platelet aggregation; Diabetic; Aspirin.
MeSH Terms: conditions — Diabetes Mellitus | interventions — Aspirin; Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pioglitazone with or without Aspirin (Experimental): Blood samples will be taken at time 0 to measure platelet aggregation. 30mg Pioglitazone will be ingested and another blood sample will be obtained 90-180 minutes later for platelet aggregation. After 6-9 days, subjects will ingest 81mg of aspirin. Another blood sample will be obtained 2-24 hours later for baseline determination of platelet aggregation and activation after taking aspirin. Subjects will then ingest 30mg pioglitazone and a final blood sample will be obtained 90-180 minutes later to measure platelet aggregation.
  Interventions: Drug: Aspirin; Drug: Pioglitazone

INTERVENTIONS:
Drug: Aspirin — 81 mg
Drug: Pioglitazone — 30mg Pioglitazone x1
  Other Names: Actos

SUMMARY:
The purpose of this study is to determine how pioglitazone and aspirin affect platelets in the blood of diabetic and non-diabetic subjects. Platelets are small cells in the blood that help with blood clotting. Pioglitazone is a drug that is used to lower blood sugar and fats by helping the body to use insulin correctly. Pioglitazone is presently used to treat diabetes but has not been approved for non-diabetics. This study will determine whether pioglitazone reduces the activity of platelets in people who are or are not also taking aspirin.

DETAILED DESCRIPTION:
Blood samples will be taken at time 0 to measure platelet aggregation. 30mg Pioglitazone will be ingested and another blood sample will be obtained 90-180 minutes later for platelet aggregation. After 6-9 days, subjects will ingest 81mg of aspirin. Another blood sample will be obtained 2-24 hours later for baseline determination of platelet aggregation and activation after taking aspirin. Subjects will then ingest 30mg pioglitazone and a final blood sample will be obtained 90-180 minutes later to measure platelet aggregation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be over 21 years of age and provide written informed consent.
* Normal subjects must have a BMI <30 and must not have known cardiovascular disease, Diabetes Mellitus (DM), hyperlipidemia, or hypertension. Diabetic subjects must have previously diagnosed DM.

Exclusion Criteria:

* Subjects will be excluded if they have hypersensitivity to aspirin or pioglitazone, or if they are receiving warfarin or heparin therapy, are pregnant, or have congestive heart failure or hepatic function impairment.
* Subjects must not have taken aspirin or other drugs inhibiting platelet function such as Plavix or non-steroidal anti-inflammatory drugs for 7 days.
* Subjects will be excluded if they have a history of renal failure, severe liver disease, myeloproliferative disease or other conditions that impair platelet function.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-12; Primary Completion 2010-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles W Francis, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

REFERENCES:
- [Derived] Mongan J, Mieszczanska HZ, Smith BH, Messing SP, Phipps RP, Francis CW. Pioglitazone inhibits platelet function and potentiates the effects of aspirin: a prospective observation study. Thromb Res. 2012 Jun;129(6):760-4. doi: 10.1016/j.thromres.2011.12.019. Epub 2012 Jan 4. PMID 22225857

RESULTS

PARTICIPANT FLOW:
Groups:
- Pioglitazone With or Without 81mg Aspirin: Blood samples will be taken at time 0 to measure platelet aggregation. 30mg Pioglitazone will be ingested and another blood sample will be obtained 90-180 minutes later for platelet aggregation. After 6-9 days, subjects will ingest 81mg of aspirin. Another blood sample will be obtained 2-24 hours later for baseline determination of platelet aggregation and activation after taking aspirin. Subjects will then ingest 30mg pioglitazone and a final blood sample will be obtained 90-180 minutes later to measure platelet aggregation.
Period: Overall Study
Arm/Group | Pioglitazone With or Without 81mg Aspirin
Started | 40
Completed | 38
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Pioglitazone With or Without 81mg Aspirin
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 34
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Percent Platelet Aggregation Induced by Arachidonic Acid
Description: Platelet aggregation was performed by the turbidimetric method of Born with simultaneous measurement of ATP release using a Chrono-log Lumi-Aggregometer with AGGRO/LINK for Windows Software version 5.1.6. Platelet rich plasma was placed in a silicone-coated cuvette with constant stirring at 1200 rpm using a siliconized stir bar for measurement of aggregation and ATP release. Aggregation was initiated using arachidonic acid (0.5 mM). At each time point the results are shown for maximum percent aggregation with arachidonic acid for all subjects. Sample 1 was obtained at baseline (BL). Sample 2 was drawn on the same day after ingestion of a single dose of 30 mg of pioglitazone. Sample 3 was obtained 6-9 days later after the subject had ingested a single 81 mg dose of aspirin (ASA), and sample 4 was drawn later that day after ingestion of 30 mg of pioglitazone.
Time Frame: at baseline and days 6-9
Population: Analysis population determined per protocol.
Measure: Mean (Standard Deviation); unit: maximum percentage aggregation
Arm/Group | Pioglitazone With or Without 81mg Aspirin
Number analyzed (Participants) | 40
maximum percentage aggregation
  Sample 1 | 80 (5)
  Sample 2 | 90 (3)
  Sample 3 | 60 (6)
  Sample 4 | 29 (6)

2. Primary Outcome: Percent Platelet Aggregation Induced by Collagen
Description: Platelet aggregation was performed by the turbidimetric method of Born with simultaneous measurement of ATP release using a Chrono-log Lumi-Aggregometer with AGGRO/LINK for Windows Software version 5.1.6. Platelet rich plasma was placed in a silicone-coated cuvette with constant stirring at 1200 rpm using a siliconized stir bar for measurement of aggregation and ATP release. Aggregation was initiated using collagen (2ug.mL). At each time point the results are shown for maximum percent aggregation with collagen for all subjects. Sample 1 was obtained at baseline (BL). Sample 2 was drawn on the same day after ingestion of a single dose of 30 mg of pioglitazone. Sample 3 was obtained 6-9 days later after the subject had ingested a single 81 mg dose of aspirin (ASA), and sample 4 was drawn later that day after ingestion of 30 mg of pioglitazone.
Time Frame: baseline and day 6-9
Measure: Mean (Standard Deviation); unit: maximum percentage aggregation
Arm/Group | Pioglitazone With or Without 81mg Aspirin
Number analyzed (Participants) | 40
maximum percentage aggregation
  Sample 1 | 89 (3)
  Sample 2 | 93 (2)
  Sample 3 | 83 (3)
  Sample 4 | 78 (3)

ADVERSE EVENTS:
Arm/Group | Pioglitazone With or Without 81mg Aspirin
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less